### INFORMED CONSENT DOCUMENT

Project Title: Residential MapTrek

Principal Investigator: Lucas Carr

**Research Team Contact:** Katie Hosteng; 319-4382221 or katie-hosteng@gmail.com

This consent form describes the research study to help you decide if you want to participate. This form provides important information about what you will be asked to do during the study, about the risks and benefits of the study, and about your rights as a research subject.

- If you have any questions about or do not understand something in this form, you should ask the research team for more information.
- You should discuss your participation with anyone you choose such as family or friends.
- Do not agree to participate in this study unless the research team has answered your questions and you decide that you want to be part of this study.

## WHAT IS THE PURPOSE OF THIS STUDY?

This is a research study. We are inviting you to participate in this research study because you are an older adult living in a residential living facility, or you are a staff member at a residential living facility. The purpose of this research study is to determine if our map-based race can encourage older adults to exercise more.

## **HOW MANY PEOPLE WILL PARTICIPATE?**

Approximately 100 people will take part in this study conducted by investigators at the University of Iowa

### **HOW LONG WILL I BE IN THIS STUDY?**

If you agree to take part in this study, your involvement will last for approximately 3 months. The initial visit will take approximately 40 minutes. For 13 weeks, you will wear the Fitbit every day. For the first eight weeks you will play our map-based racing game, MapTrek. For the last four weeks, you will only wear the Fitbit. Once you are done playing MapTrek, we will collect some additional survey data from you that will take about 10-15 minutes to collect.

### WHAT WILL HAPPEN DURING THIS STUDY?

We will first ask you to fill out a brief activity survey interview style. We will ask you for some basic demographic information such as your age, gender, and race/ethnicity. We will also ask you questions about physical activity. You are free to skip any questions that you prefer not to answer. We will then ask you to wear a Fitbit for 24 hours a day (except during bathing or swimming) so that we may collect baseline data from you for 4 days. The Fitbit will collect activity measurements (i.e., steps and minutes of physical activity per day) in 1-minute intervals throughout the entire study.

After the baseline period, you will be placed onto one of three possible teams, based on your baseline physical activity data. Teams will stay the same throughout the study and will be designated by different colored Fitbit bands (black, white or teal). The three teams will compete against each other in walking 'races' for the next eight weeks using MapTrek. MapTrek is a web-based application that allows users

Page 2 of 5

to take a virtual walk in interesting locations around the world while tracking their progress against the progress of others who are also playing. Each race will open on a Monday morning and the winners and final standings will be declared on the Sunday two weeks after the race begins. You will be asked to participate in four different races over the course of 8 weeks.

Each day, we will ask you to walk by a TV monitor or other syncing stations in your residential living facility to sync your Fitbit, view physical activity information for your team, and view the leaderboard. The monitors will only present aggregated team data and will not report any of your own individual data.

At the end of the 8-weeks of walking races, we will ask you to complete an exit survey. The survey will ask you about physical activity as well as your thoughts and opinions of the MapTrek game. We will collect the survey responses from you via phone or in person (whichever you prefer). This survey should take about 10-15 minutes to complete. We will also ask you if you would like to participate in a focus group at the end of the 8-weeks of walking races. During the focus group we will ask you questions about what you liked and disliked about the game, as well as any suggestions you have for future studies. The focus groups will be audio recorded with a digital recorder.

We will then ask you to wear the Fitbit for an additional four weeks without playing the MapTrek game. We will continue collecting activity measurements (i.e., steps and minutes of physical activity per day) in 1-minute intervals for four more weeks. We will ask you to continue syncing your Fitbit during this time at the syncing stations. Once the four-week data collection period is over we will let you know that you are done with the study.

# **Data Storage for Future Use**

As part of this study, we are obtaining physical activity data from you. We would like to study your physical activity data in the future, after this study is over.

The tests we might want to use to study your data may not even exist at this time. Therefore, we are asking for your permission to store your data so that we can study them in the future. These future studies may provide additional information that will help in understanding how to increase physical activity in older adults, but it is unlikely that what we learn from these studies will have a direct benefit to you. It is possible that your data might be used to develop products or tests that could be patented and licensed. There are no plans to provide financial compensation to you should this occur.

Your physical activity data will be stored with a code which may be linked to your name and phone number. If you agree now to future use of your physical activity data but decide in the future that you would like to have it removed from future research, you should contact **Dr. Lucas Carr, PhD at 319-353-5432**. However, if some research with your physical activity data has already been completed, the information from that research may still be used.

Please place your initials in the blank next to Yes or No below:

| My data may be stored for future research for any other purpose. | |
|------------------------------------------------------------------|----|
| Yes | No |

## WHAT ARE THE RISKS OF THIS STUDY?

You might feel tired or may possibly be injured as a result of being more physically active than usual. To minimize this risk the intervention will only promote engagement in low to moderate intensity physical activity which poses a low risk for injury. In addition to this, there may be other unknown risks, or risks that we did not anticipate, associated with being in this study.

### WHAT ARE THE BENEFITS OF THIS STUDY?

You will not benefit from being in this study. However, we hope that, in the future, other people might benefit from this study because of knowledge gained in determining if competition will encourage older adults living in a retirement community to exercise more.

# WILL IT COST ME ANYTHING TO BE IN THIS STUDY?

You will not have any costs for being in this research study.

### WILL I BE PAID FOR PARTICIPATING?

All participants will be able to keep the Fitbit activity monitor at the end of the study.

Participants who attend a focus group session will receive a \$50 check in the mail. You will need to provide your name and address in order to have the check issued.

## WHO IS FUNDING THIS STUDY?

The University and the research team are receiving no payments from other agencies, organizations, or companies to conduct this research study.

# WHAT ABOUT CONFIDENTIALITY?

We will keep your participation in this research study confidential to the extent permitted by law. However, it is possible that other people such as those indicated below may become aware of your participation in this study and may inspect and copy records pertaining to this research. Some of these records could contain information that personally identifies you.

- federal government regulatory agencies,
- auditing departments of the University of Iowa, and
- the University of Iowa Institutional Review Board (a committee that reviews and approves research studies)

To help protect your confidentiality, we will assign a study ID to your data instead of using your name. The study ID will be linked to your name. The list linking your name and your study identification code will be stored in a separate location that is accessible only to the researchers. We will store all of the data we collect from you on a secure server that can only be accessed by the research team. Paper forms will be kept in a locked cabinet in a locked office. If we write a report or article about this study or share the study data set with others, we will do so in such a way that you cannot be directly identified.

### IS BEING IN THIS STUDY VOLUNTARY?

Taking part in this research study is completely voluntary. You may choose not to take part at all. If you decide to be in this study, you may stop participating at any time. If you decide not to be in this study, or if you stop participating at any time, you won't be penalized or lose any benefits for which you

otherwise qualify.

### What if I Decide to Drop Out of the Study?

If you decide to leave the study early, we will ask you to contact **Katie Hosteng at 319-438-2221** or **katie-hosteng@uiowa.edu**.

## WHAT IF I HAVE QUESTIONS?

We encourage you to ask questions. If you have any questions about the research study itself or if you experience a research-related injury, please contact **Katie Hosteng at 319-438-2221** or <a href="mailto:katie-hosteng@uiowa.edu">katie-hosteng@uiowa.edu</a>.

If you have questions, concerns, or complaints about your rights as a research subject or about research related injury, please contact the Human Subjects Office, 105 Hardin Library for the Health Sciences, 600 Newton Rd, The University of Iowa, Iowa City, IA 52242-1098, (319) 335-6564, or e-mail <a href="mailto:irb@uiowa.edu">irb@uiowa.edu</a>. General information about being a research subject can be found by clicking "Info for Public" on the Human Subjects Office web site, <a href="http://hso.research.uiowa.edu/">http://hso.research.uiowa.edu/</a>. To offer input about your experiences as a research subject or to speak to someone other than the research staff, call the Human Subjects Office at the number above.

This Informed Consent Document is not a contract. It is a written explanation of what will happen during the study if you decide to participate. You are not waiving any legal rights by signing this Informed Consent Document. Your signature indicates that this research study has been explained to you, that your questions have been answered, and that you agree to take part in this study. You will receive a copy of this form.

| Subject's Name (printed): | |
|---|---|
| Do not sign this form if today's date is on | or after EXPIRATION DATE: 05/29/21. |
| (Signature of Subject) | (Date) |
| Statement of Person Who Obtained Conse | <u>ent</u> |
| <u> </u> | ubject or, where appropriate, with the subject's legally that the subject understands the risks, benefits, and is research study. |
| (Signature of Person who Obtained Consent | (Date) |